CLINICAL TRIAL: NCT05337631
Title: Special Care Patterns for Elderly HNSCC Patients Undergoing Radiotherapy
Acronym: SENIOR
Status: Recruiting | Type: Observational
Sponsor: University Hospital Freiburg (Other)
Collaborators: Charite University, Berlin, Germany (Other); Johann Wolfgang Goethe University Hospital (Other); University Hospital, Zürich (Other); Wuerzburg University Hospital (Other); University Hospital Schleswig-Holstein (Other); Johannes Gutenberg University Mainz (Other); University Hospital Munich (Other); Friedrich-Alexander-Universität Erlangen-Nürnberg (Other); Case Western Reserve University (Other); Icahn School of Medicine at Mount Sinai (Other); Ohio State University (Other); German Oncology Center, Cyprus (Other); University of Leipzig (Other); Johns Hopkins University (Other); Martin-Luther-Universität Halle-Wittenberg (Other); University of Giessen (Other); Brno University Hospital (Other); Jena University Hospital (Other)
Responsible Party: Principal Investigator, Nils Nicolay, Professor and Vice Chair, Department of Radiation Oncology, University Hospital Freiburg
Other Study IDs: FRKS003723
Record Dates: First submitted 2022-03-07; First posted 2022-04-20 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: HNSCC; Oral Cavity Cancer; Oropharynx Cancer; Hypopharynx Cancer; Larynx Cancer
Keywords: Elderly; Radiotherapy; Chemotherapy; Chemoradiotherapy; Cisplatin; Cetuximab; Real-world data
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Mouth Neoplasms; Oropharyngeal Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The number of elderly head-and-neck squamous cell carcinoma (HNSCC) patients is increasing; however, the evidence regarding the ideal treatment for this often vulnerable and frail patient cohort is limited. Although the benefit of concomitant chemotherapy has been reported to decrease in elderly HNSCC patients based on the MACH-NC meta-analysis, it remains unknown whether state-of-the art radiotherapy techniques such as intensity-modulated radiotherapy (IMRT), modern supportive treatments and alternative chemotherapy fractionation (e.g., cisplatin weekly) may have altered this observation. The objective of this retrospective multinational multicenter study is to determine the oncological outcomes of elderly patients (≥65 years) with locally advanced HNSCCs undergoing definitive (chemo-)radiation and to investigate the influence of concomitant chemotherapy on overall survival and progression-free survival after adjusting for potential confounder variables such as age, performance status and comorbidity burden.

ELIGIBILITY:
Inclusion Criteria:

* definitive (chemo-)radiotherapy of locoregionally advanced (cT3-4 and/or cN+) head-and-neck squamous cell carcinomas (HNSCC) of the oral cavity, oropharynx, hypopharynx or larynx
* primary treatment since 2005
* age ≥65 years at the time of (chemo-)radiotherapy

Exclusion Criteria:

* adjuvant (chemo-)radiotherapy
* history of previous head-and-neck cancers or radiotherapy in the head-and-neck region
* distant metastases at (chemo-)radiotherapy initiation (cM1)
* HNSCCs of the nasopharynx, salivary glands, skin or with unknown primary

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly (≥65 years) head-and-neck squamous cell carcinoma (HNSCC) patients undergoing definitive (chemo)radiotherapy since 2005 at a tertiary cancer center will be included and analyzed in terms of overall survival and the potential benefit of concomitant chemotherapy administration.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to 5 years
  Time from radiotherapy start until death from any cause

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 5 years
  Time from radiotherapy start until death from any cause, local progression, locoregional progression or distant progression (whichever occurs first)

OTHER OUTCOMES:
Patterns of chemotherapy administration | during radiotherapy
  Type of concomitant chemotherapy
Cumulative cisplatin dose | during radiotherapy
  Dose of concomitant cisplatin in mg/m2 body surface area
Radiotherapy compliance | during treatment
  Radiotherapy completion rate
Chemotherapy compliance | during treatment
  Chemotherapy completion rate

CONTACTS AND LOCATIONS:
Overall Officials: Nils H. Nicolay, MD, PhD, Principal Investigator — Department of Radiation Oncology, Medical Center - University of Freiburg; Alexander Rühle, MD, Principal Investigator — Department of Radiation Oncology, Medical Center - University of Freiburg
Locations (18):
- United States (4):
  - Department of Radiation Oncology and Molecular Radiation Sciences, Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Department of Radiation Oncology, Icahn School of Medicine at Mount Sinai, New York, New York
  - Department of Radiation Oncology, Case Western Reserve University, Cleveland, Ohio
  - Division of Radiation Oncology, The Ohio State University Wexner, Columbus, Ohio
- Radiation Oncology Department, German Oncology Center, Limassol, Cyprus
- Brno University Hospital, Brno, Czechia
- Germany (11):
  - Department of Radiooncology and Radiotherapy, Charité-Universitätsmedizin Berlin, Berlin
  - Department of Radiation Oncology, University Hospital Erlangen, Friedrich-Alexander-University Erlangen-Nürnberg, Erlangen
  - Department of Radiotherapy and Oncology, Goethe-University Frankfurt am Main, Frankfurt
  - University of Giessen, Giessen
  - Martin-Luther-Universität Halle-Wittenberg, Halle
  - Jena University Hospital, Jena
  - Department of Radiation Oncology, University Hospital Schleswig-Holstein, Kiel
  - Department of Radiation Oncology, University Medical Center Leipzig, Leipzig
  - Department of Radiation Oncology, University Medical Center Mainz, Mainz
  - Department of Radiation Oncology, University Hospital, LMU Munich, Munich
  - Department of Radiation Oncology, University Hospital Würzburg, Würzburg
- Department of Radiation Oncology, University Hospital Zurich (USZ), University of Zurich (UZH), Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2024-07-26): https://cdn.clinicaltrials.gov/large-docs/31/NCT05337631/Prot_001.pdf